CLINICAL TRIAL: NCT04039139
Title: Mind Body Therapy for the Treatment of Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Michael Donnino, Associate Professor of Emergency Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018P000578
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Chronic Pain; Chronic Pain Syndrome
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Usual Care, Intervention
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be partially blinded. Participants in the usual care arm will be blinded to the specifics of the interventions. Intervention participants will be blinded to the specifics of the intervention until after they have been randomized into that arm. Data analysis will be conducted by persons who are completely blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): Participants will continue their usual care for 26 weeks
- Mind Body Intervention 1: Mind-Body-Syndrome-Therapy (MBST) (Experimental): Participants will receive a mind body educational-based intervention to learn the techniques comprising intervention 1. Further details are not provided for blinding purposes.
  Interventions: Behavioral: Mind Body Intervention 1: Mind-Body-Syndrome-Therapy (MBST)
- Mind Body Intervention 2 (Active Comparator): Participants will receive a mind-body educational-based intervention to learn the techniques comprising intervention 2. Further details are not provided for blinding purposes.
  Interventions: Behavioral: Mind Body Intervention 2

INTERVENTIONS:
Behavioral: Mind Body Intervention 1: Mind-Body-Syndrome-Therapy (MBST) — Mind body techniques for Intervention 1 will be taught in lectures and group discussion sessions.
  Other Names: MBST
  Arms: Mind Body Intervention 1: Mind-Body-Syndrome-Therapy (MBST)
Behavioral: Mind Body Intervention 2 — Mind body techniques for Intervention 2 will be taught in lectures and group and/or individual sessions.
  Arms: Mind Body Intervention 2

SUMMARY:
Chronic pain syndromes without identified organic etiology remain a challenge for physicians. Many syndromes, including back pain, are believed to have potential underlying psychological etiology; however, the exact link remains elusive. The goal of this study is to determine if mind body therapies can help people suffering from chronic back pain. The study is a randomized, partially blinded trial examining the effectiveness of Mind Body Syndrome Therapy (MBST) in reducing disability from back pain and alleviating back pain. The investigators will secondarily investigate whether MBST can improve participant quality of life and reduce the need for pain-related hospitalization. The design of the this study consists of 3 arms with one being the intervention (MBST), one being usual care, and one being a second mind-body intervention (active control). This education program consists of a series of personal interviews and group and/or individualized lectures/sessions. Participants will also be provided reading material to study during the intervention period, and asked to continue their usual care while going through the MBST program.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient 18 > years old
* Chronic back pain
* Pain persistent for ≥3 days/week for the past 3 months prior to enrollment
* Willingness to consider mind-body intervention

Exclusion Criteria:

* Patients < 18 years of age
* Diagnosed organic disease as cause of pain, such as (but not limited) to malignancy, neurologic disorder (i.e., amyotrophic lateral sclerosis), cauda equina syndrome. Pain related to disc disease is not an exclusion unless there are neurological impairments.
* Patients with a diagnosis of significant psychiatric co-morbidities such as schizophrenia, dementia and bipolar disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Pain Disability: Roland Morris Disability Index | change over 26 weeks
  Change in the Roland Morris Disability Index (Scale 0-24 with 24 being worst)

SECONDARY OUTCOMES:
Average Pain: Brief Pain Inventory Survey | 4 weeks, 8 weeks, 13, weeks, 26 weeks
  Average pain as determined in the Brief Pain Inventory Survey (Scale 0-10 with 10 being worst)
Pain Bothersomeness (Back Specific): Brief Pain Inventory Survey | 4 weeks, 8 weeks, 13 weeks, 26 weeks
  Back pain bothersomeness as determined from modified Brief Pain Inventory Survey. (Scale 0-10 with 10 being the worst)
Pain Bothersomeness: Brief Pain Inventory Survey | 4 weeks, 8 weeks, 13 weeks, 26 weeks
  Whole-body pain bothersomeness as determined from modified Brief Pain Inventory Survey (Scale of 0-10 with 10 being the worst)
Pain affecting enjoyment of life | 4 weeks, 8 weeks, 13 weeks, 26 weeks
  Scale 0-10 with 10 being worst from Brief Pain Inventory
Anxiety from pain: Pain Anxiety Symptom Scale-20 survey | 4 weeks, 8 weeks, 13 weeks, 26 weeks
  Anxiety from pain as determined from the Pain Anxiety Symptom Scale-20 survey (20 questions with scale of 0-5 with 5 being 'always' and 0 being 'never'
Pain-related hospital admissions | 26 weeks
  Self reported. Number of pain-related hospital admissions, including emergency room visits
Complete resolution of pain disability: Roland Morris Disability | 4 weeks, 8 weeks, 13 weeks, 26 weeks
  complete resolution of pain disability as measured by Roland Morris Disability (Scale 0-24 with 24 being worst)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Donnino, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
The investigators will not be sharing IPD data with researchers outside of their research group.